CLINICAL TRIAL: NCT04781777
Title: Effect of Ultrasonographic Guided Insulin Injection With Dexamethasone and Local Anesthetic Mixture in Diabetic Patients With Mild to Moderate Carpal Tunnel .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124/2-2021.
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Pain Relief
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Dexmehtasone and local anesthetics in carpal tunnel syndrome
- Insulin group (Active Comparator): insulin added to dexamehtasone and local anesthetics
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — sonar guided insulin combined with dexamethasone and local anesthetics
  Other Names: Sonar guided median nerve hydrodissection
  Arms: Insulin group

SUMMARY:
Insulin as an adjuvant to local anesthetic and cortisone to decrease pain recurrence

ELIGIBILITY:
Inclusion Criteria:

- Diabetic patients with mild to moderate carpal tunnel syndrome

Exclusion Criteria:

* Refusal to participate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
pain neuropathy | 12 weeks
  relief chronic pain from caroal tunnel